CLINICAL TRIAL: NCT01065298
Title: Efficacy Of Autologous Bone Marrow Derived Stem Cell Transplantation In Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy Of Autologous Bone Marrow Derived Stem Cell Transplantation In Patients With Type 2 Diabetes Mellitus-2
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, head of department, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: ABMSCT2
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1:Stem cell Recipient: Patients with Type 2 Diabetes mellitus on full doses of Vildagliptin+Pioglitazone+Metformin and requiring Insulin at dose of >0.4U/Kg for blood glucose control. They will undergo stem cell therapy initialy and G-CSF therapy at 2 months
  Interventions: Biological: stem cell transplantation
- Group-2: Controls: Type 2 Diabetes mellitus patients on full doses of vildagliptin+metformin+pioglitazone and on Insulin >0.4U/Kg who will act as active control.They will receive injectable placebo at Day 1 in addition to above and will be followed up for 6 months.Follow up investigation and Insulin dose titration will be similar to Group 1.

INTERVENTIONS:
Biological: stem cell transplantation — Group 1: 200 - 250 ml of bone marrow will be aspirated and layered on density gradient medium (Ficoll - Hyperaque) and stem cells will be separated. Separated MNC's will be tagged with FDG-PET and injected into superior pancreatico duodenal artery and an PET scan will be done 2 hours later to see the percentage of stem cells homing in to pancreas. After 8 weeks G-CSF(10mcg/Kg/day) will be given subcutaneous for 5 days to achieve a Leucocyte count of >40,000/mm3. Patients will be urged to monitor and document blood glucose readings for next 6 months. Glucagon stimulated C - peptide, plasma Insulin, HOMA-IR , HOMA-B ,HbA1c, lipid profile and biochemistry will be done at baseline and 6 months .
  Other Names: Autologous Bone marrow derived stem cell transplantation
  Groups: Group 1:Stem cell Recipient

SUMMARY:
The purpose of this study is to improve blood glucose control in Type 2 Diabetes mellitus patients.

DETAILED DESCRIPTION:
We hypothesize that Autologous bone marrow derived stem cell transplantation(ABMSCT)into the pancreas of patients with T2DM, aged 30 - 70 years with triple oral hypoglycemic agent failure and on insulin(>0.4 U/ kg body weight/day) will lead to abolition or reduction of insulin requirement by more than or equal to 50% in these patients over a period of 6 months. It is assumed that ABMSCT in these patients leads to increased angiogenesis, secretion of various cytokines and upregulation of pancreatic transcription factors and Vascular endothelial growth factor(VEGF) and creates a microenvironment which supports beta cell/resident stem cell activation and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus between 30 and 70 years of age.
2. Failure to triple OHA and on stable doses of insulin for atleast 3 months.
3. On vildagliptin,pioglitazone and metformin for atleast 3 months along with Insulin to maintain euglycemia.
4. HbA1c < 8.5%.
5. Insulin requirement ≥0.4 IU/kg/d.
6. GAD antibody negative status.

Exclusion Criteria:

1. Patients with T1DM or secondary diabetes.
2. Patients with serum creatinine > 1.5 mg/dl.
3. Abnormal liver function tests (defined as value of transaminases > 3 times the upper value of normal or serum bilirubin higher than normal for the reference value for the laboratory).
4. History of cholecystitis/ cholelitiasis/ cholecystectomy
5. Seropositivity for HIV, HBsAg and HCV.
6. History of myocardial infarction or unstable angina in the previous 3 months.
7. History of malignancy
8. Patients with active infections.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 Diabetes mellitus with triple Oral hypoglycemic failure and on Insulin for glycemic control
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Reduction of insulin requirement by ≥ 50% by the end of 6 months of ABMSCT and Improvement in Glucagon stimulated C - peptide levels . | 6 months

SECONDARY OUTCOMES:
Any reduction in requirement of insulin dosage and any improvement of HbA1c levels as compared to controls. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, MD.,DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; Neelam Marwaha, MD.,DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; N Khandelwal, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; B.R. Mittal, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Prem Kumar, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Rama Walia, MD.,DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh UT, India

REFERENCES:
- [Result] Bhansali A, Upreti V, Khandelwal N, Marwaha N, Gupta V, Sachdeva N, Sharma RR, Saluja K, Dutta P, Walia R, Minz R, Bhadada S, Das S, Ramakrishnan S. Efficacy of autologous bone marrow-derived stem cell transplantation in patients with type 2 diabetes mellitus. Stem Cells Dev. 2009 Dec;18(10):1407-16. doi: 10.1089/scd.2009.0164. PMID 19686048